CLINICAL TRIAL: NCT01848834
Title: A Phase Ib Multi-Cohort Study of MK-3475 in Subjects With Advanced Solid Tumors
Brief Title: Study of Pembrolizumab (MK-3475) in Participants With Advanced Solid Tumors (MK-3475-012/KEYNOTE-012)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-012; 2012-005771-14 (EudraCT Number); 142453 (Registry Identifier: JAPIC_CTI); MK-3475-012 (Other: Merck)
Record Dates: First submitted 2013-05-03; First posted 2013-05-08 (Estimated); Results first posted 2017-06-26 (Actual); Last update posted 2021-06-28 (Actual); Status verified 2021-05

CONDITIONS: Cancer; Solid Tumor
Keywords: PD-1; PD1; PD-L1; PDL1
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort A: Triple Negative Breast Cancer (Experimental): Participants receive pembrolizumab, 10 mg/kg, intravenously (IV) once every 2 weeks, and continue to receive drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years).
  Interventions: Biological: Pembrolizumab
- Cohort B: Head & Neck Cancer (Experimental): Participants receive pembrolizumab, 10 mg/kg, IV once every 2 weeks, and continue to receive drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years).
  Interventions: Biological: Pembrolizumab
- Cohort C: Urothelial Cancer (Experimental): Participants receive pembrolizumab, 10 mg/kg, IV once every 2 weeks, and continue to receive drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years).
  Interventions: Biological: Pembrolizumab
- Cohort D: Gastric Cancer (Experimental): Participants receive pembrolizumab, 10 mg/kg, IV once every 2 weeks, and continue to receive drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years).
  Interventions: Biological: Pembrolizumab
- Cohort B2: Head & Neck Cancer Expansion (Experimental): Participants receive pembrolizumab, 200 mg, IV once every 3 weeks, and continue to receive drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years).
  Interventions: Biological: Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; SCH 900475; KEYTRUDA®

SUMMARY:
This study is being done to investigate the safety, tolerability and anti-tumor activity of pembrolizumab (MK-3475) in participants with advanced triple negative breast cancer (TNBC) (Cohort A), advanced head and neck cancer (Cohorts B and B2), advanced urothelial cancer (Cohort C), or advanced gastric cancer (Cohort D). Additionally, for Cohort D, data is presented for Asian Pacific (AP) participants. Only participants with programmed cell death-ligand 1 (PD-L1) expressing tumors were enrolled in Cohorts A, B, C and D. Participants in Cohort B2 were enrolled irrespective of PD-L1 status.

The primary study hypothesis is that pembrolizumab is safe and well-tolerated.

DETAILED DESCRIPTION:
Eligible participants who completed the first course of up to 35 administrations of pembrolizumab (approximately up to 2 years) for reasons other than disease progression or intolerability, may be eligible for a second course of pembrolizumab for up to approximately 1 additional year at the investigator's discretion. Per protocol, response during this second course will not count towards the efficacy outcome measures and adverse events during this second course will not count towards the safety outcome measures.

Protocol Amendment 01 (08 Aug 2013) included a new study arm (Cohort D) for approximately 32 participants with advanced gastric cancer. Of these 32 participants, 16 will be from sites in the Asia Pacific (AP) region and the other 16 will be from sites outside the AP region.

Protocol Amendment 02 (07 Apr 2014) added a new study arm (Cohort B2) for approximately 110 participants with advanced head and neck cancer who will receive a lower dose of pembrolizumab every three weeks (Q3W). Both programmed cell death ligand 1 (PD-L1)- positive and PD-L1-negative participants will be enrolled into this cohort.

Protocol Amendment 03 (26 May 2015) removed the secondary objective of investigating the relationship between programmed cell death 1 (PD-1) inhibition and up-regulation of cytokines biomarkers predicting response (e.g. Interleukin-10 [IL-10]) from the protocol.

Participants who stopped study treatment without progression (e.g. completed 2 years) may have been eligible for up to 1 year of retreatment upon subsequently experiencing disease progression.

With Amendment 05 (11 Dec 2017), once study participants have achieved the study objective or the study has ended, participants will be discontinued from this study and enrolled in an extension study (KEYNOTE-587; NCT03486873) to continue protocol-defined assessments and treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed diagnosis of tumor that is recurrent, metastatic, or persistent:

  * For Cohort A - triple negative breast cancer (estrogen, progesterone, and human epidermal growth factor receptor 2 [HER2] negative)
  * For Cohort B - squamous cell carcinoma of the head and neck (including human papilloma virus (HPV)-positive head and neck squamous cell cancer).
  * For Cohort C - urothelial tract cancer of the renal pelvis, ureter, bladder, or urethra (transitional cell or non-transitional cell histology)
  * For Cohort D - adenocarcinoma of the stomach or gastroesophageal junction
  * For Cohort B2 - squamous cell carcinoma of the head and neck (both HPV-positive and -negative head and neck squamous cell cancer)
* Any number of prior treatment regimens
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0 or 1
* Female participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study treatment
* Male participants must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study treatment

Exclusion Criteria:

* Currently participating in/has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study treatment
* Diagnosis of immunosuppression or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Anti-cancer monoclonal antibody treatment within 4 weeks prior to study Day 1 or not recovered from adverse events due to agents administered more than 4 weeks earlier
* Chemotherapy, targeted small molecule therapy or radiation therapy within 2 weeks prior to study Day 1 or not recovered from adverse events due to a previously administered agent
* Known additional malignancy that is progressing or requires active treatment excepting basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease requiring systemic treatment within the past 3 months or documented history of clinically severe autoimmune disease, or syndrome that requires systemic steroids or immunosuppressive agents
* Evidence of interstitial lung disease
* Active infection requiring systemic therapy
* Known psychiatric or substance abuse disorders
* Pregnant, breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Prior therapy with an anti-programmed cell death 1 (PD-1), anti-PD-L1, anti-PD-L2, anti-CD137 antibody, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody
* Known history of human immunodeficiency virus (HIV)
* Known active Hepatitis B or Hepatitis C
* Received live vaccine within 30 days prior to start of study treatment
* Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is Investigational site or Sponsor staff directly involved with this trial, unless prospective Independent Review Board (IRB) approval (by Chair or Designee) is given allowing exception to this criterion for a specific participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Actual)
Dates: Start 2013-05-07 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Muro K, Chung HC, Shankaran V, Geva R, Catenacci D, Gupta S, Eder JP, Golan T, Le DT, Burtness B, McRee AJ, Lin CC, Pathiraja K, Lunceford J, Emancipator K, Juco J, Koshiji M, Bang YJ. Pembrolizumab for patients with PD-L1-positive advanced gastric cancer (KEYNOTE-012): a multicentre, open-label, phase 1b trial. Lancet Oncol. 2016 Jun;17(6):717-726. doi: 10.1016/S1470-2045(16)00175-3. Epub 2016 May 3. PMID 27157491
- [Result] Nanda R, Chow LQ, Dees EC, Berger R, Gupta S, Geva R, Pusztai L, Pathiraja K, Aktan G, Cheng JD, Karantza V, Buisseret L. Pembrolizumab in Patients With Advanced Triple-Negative Breast Cancer: Phase Ib KEYNOTE-012 Study. J Clin Oncol. 2016 Jul 20;34(21):2460-7. doi: 10.1200/JCO.2015.64.8931. Epub 2016 May 2. PMID 27138582
- [Result] Seiwert TY, Burtness B, Mehra R, Weiss J, Berger R, Eder JP, Heath K, McClanahan T, Lunceford J, Gause C, Cheng JD, Chow LQ. Safety and clinical activity of pembrolizumab for treatment of recurrent or metastatic squamous cell carcinoma of the head and neck (KEYNOTE-012): an open-label, multicentre, phase 1b trial. Lancet Oncol. 2016 Jul;17(7):956-965. doi: 10.1016/S1470-2045(16)30066-3. Epub 2016 May 27. PMID 27247226
- [Result] Plimack ER, Bellmunt J, Gupta S, Berger R, Chow LQ, Juco J, Lunceford J, Saraf S, Perini RF, O'Donnell PH. Safety and activity of pembrolizumab in patients with locally advanced or metastatic urothelial cancer (KEYNOTE-012): a non-randomised, open-label, phase 1b study. Lancet Oncol. 2017 Feb;18(2):212-220. doi: 10.1016/S1470-2045(17)30007-4. Epub 2017 Jan 10. PMID 28081914
- [Result] Chow LQM, Haddad R, Gupta S, Mahipal A, Mehra R, Tahara M, Berger R, Eder JP, Burtness B, Lee SH, Keam B, Kang H, Muro K, Weiss J, Geva R, Lin CC, Chung HC, Meister A, Dolled-Filhart M, Pathiraja K, Cheng JD, Seiwert TY. Antitumor Activity of Pembrolizumab in Biomarker-Unselected Patients With Recurrent and/or Metastatic Head and Neck Squamous Cell Carcinoma: Results From the Phase Ib KEYNOTE-012 Expansion Cohort. J Clin Oncol. 2016 Nov 10;34(32):3838-3845. doi: 10.1200/JCO.2016.68.1478. Epub 2016 Sep 30. PMID 27646946
- [Derived] Haddad RI, Seiwert TY, Chow LQM, Gupta S, Weiss J, Gluck I, Eder JP, Burtness B, Tahara M, Keam B, Kang H, Muro K, Albright A, Mogg R, Ayers M, Huang L, Lunceford J, Cristescu R, Cheng J, Mehra R. Influence of tumor mutational burden, inflammatory gene expression profile, and PD-L1 expression on response to pembrolizumab in head and neck squamous cell carcinoma. J Immunother Cancer. 2022 Feb;10(2):e003026. doi: 10.1136/jitc-2021-003026. PMID 35217573
- [Derived] Cristescu R, Aurora-Garg D, Albright A, Xu L, Liu XQ, Loboda A, Lang L, Jin F, Rubin EH, Snyder A, Lunceford J. Tumor mutational burden predicts the efficacy of pembrolizumab monotherapy: a pan-tumor retrospective analysis of participants with advanced solid tumors. J Immunother Cancer. 2022 Jan;10(1):e003091. doi: 10.1136/jitc-2021-003091. PMID 35101941
- [Derived] van Vugt MJH, Stone JA, De Greef RHJMM, Snyder ES, Lipka L, Turner DC, Chain A, Lala M, Li M, Robey SH, Kondic AG, De Alwis D, Mayawala K, Jain L, Freshwater T. Immunogenicity of pembrolizumab in patients with advanced tumors. J Immunother Cancer. 2019 Aug 8;7(1):212. doi: 10.1186/s40425-019-0663-4. PMID 31395089
- [Derived] Tahara M, Muro K, Hasegawa Y, Chung HC, Lin CC, Keam B, Takahashi K, Cheng JD, Bang YJ. Pembrolizumab in Asia-Pacific patients with advanced head and neck squamous cell carcinoma: Analyses from KEYNOTE-012. Cancer Sci. 2018 Mar;109(3):771-776. doi: 10.1111/cas.13480. Epub 2018 Feb 8. PMID 29284202

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All allocated participants through end of trial (EOT) analysis cutoff date of 30 June 2020.
Groups:
- Cohort A: Triple Negative Breast Cancer: Participants received pembrolizumab, 10 mg/kg, intravenously (IV) once every 2 weeks, and continued to receive study drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years). Participants who stopped study treatment without progression (e.g. completed 2 years) may have been eligible for up to 1 year of retreatment upon subsequently experiencing disease progression.
- Cohort B: Head & Neck Cancer; Cohort C: Urothelial Cancer; Cohort D: Gastric Cancer: Participants received pembrolizumab, 10 mg/kg, IV once every 2 weeks, and continued to receive study drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years). Participants who stopped study treatment without progression (e.g. completed 2 years) may have been eligible for up to 1 year of retreatment upon subsequently experiencing disease progression.
- Cohort B2: Head & Neck Cancer Expansion: Participants received pembrolizumab, 200 mg, IV once every 3 weeks, and continued to receive study drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years). Participants who stopped study treatment without progression (e.g. completed 2 years) may have been eligible for up to 1 year of retreatment upon subsequently experiencing disease progression.
Period: Overall Study
Arm/Group | Cohort A: Triple Negative Breast Cancer | Cohort B: Head & Neck Cancer | Cohort C: Urothelial Cancer | Cohort D: Gastric Cancer | Cohort B2: Head & Neck Cancer Expansion
Started | 32 | 61 | 33 | 39 | 132
Treated | 32 | 60 | 33 | 39 | 132
Completed | 13 (Completed means two-year treatment completed) | 13 (Completed means two-year treatment completed) | 9 (Completed means two-year treatment completed) | 13 (Completed means two-year treatment completed) | 38 (Completed means two-year treatment completed)
Not Completed | 19 | 48 | 24 | 26 | 94
Not completed — Adverse Event | 3 | 11 | 3 | 5 | 9
Not completed — Death | 2 | 11 | 1 | 8 | 27
Not completed — Excluded Medication | 5 | 4 | 3 | 6 | 6
Not completed — Lost to Follow-up | 5 | 5 | 3 | 0 | 3
Not completed — Physician Decision | 1 | 3 | 4 | 0 | 11
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Sponsor Decision | 1 | 1 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 13 | 10 | 6 | 36

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all allocated participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A: Triple Negative Breast Cancer | Cohort B: Head & Neck Cancer | Cohort C: Urothelial Cancer | Cohort D: Gastric Cancer | Cohort B2: Head & Neck Cancer Expansion | Total
Number analyzed (Participants) | 32 | 61 | 33 | 39 | 132 | 297
Age, Continuous [Mean (Standard Deviation); unit: Years] | 51.9 (12.1) | 61.5 (11.5) | 68.5 (10.3) | 58.3 (13.2) | 58.9 (9.7) | 59.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 12 | 10 | 11 | 22 | 87
  Male | 0 | 49 | 23 | 28 | 110 | 210
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 1 | 1 | 7 | 12
  Not Hispanic or Latino | 29 | 58 | 23 | 37 | 108 | 255
  Unknown or Not Reported | 1 | 2 | 9 | 1 | 17 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1 | 2
  Asian | 0 | 1 | 0 | 19 | 28 | 48
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 7 | 6 | 2 | 0 | 4 | 19
  White | 25 | 53 | 31 | 19 | 95 | 223
  More than one race | 0 | 1 | 0 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 3 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. The number of participants who experienced at least one AE was presented for the first course pembrolizumab treatment per protocol.
Time Frame: Serious AEs: Up to 90 days after last dose of treatment (Up to 28 months); nonserious AEs: Up to 30 days after last dose of treatment (Up to 26 months) - through final analysis (FA) cutoff date 26 Apr 2016 (Cohorts: A, B, B2, D) & 01 Sep 2015 (Cohort C)
Population: The population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer | Cohort B: Head & Neck Cancer | Cohort C: Urothelial Cancer | Cohort D: Gastric Cancer | Cohort B2: Head & Neck Cancer Expansion
Number analyzed (Participants) | 32 | 60 | 33 | 39 | 132
Participants | 32 | 58 | 33 | 39 | 130

2. Primary Outcome: Number of Participants Discontinuing From Study Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a study treatment which did not necessarily have to have a causal relationship with this treatment. An AE could be any unfavourable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that was temporally associated with the use of study treatment, was also an AE. Some cases of clinical progression that led to discontinuation of study treatment were captured as AEs that led to discontinuation of study treatment. The number of participants who discontinued study treatment due to an AE was presented for the first course pembrolizumab treatment per protocol.
Time Frame: Up to last dose of study treatment (Up to approximately 25 months) - through FA cutoff date 26 Apr 2016 (Cohorts: A, B, B2, D) & 01 Sep 2015 (Cohort C)
Population: The population consisted of all participants who received ≥1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer | Cohort B: Head & Neck Cancer | Cohort C: Urothelial Cancer | Cohort D: Gastric Cancer | Cohort B2: Head & Neck Cancer Expansion
Number analyzed (Participants) | 32 | 60 | 33 | 39 | 132
Participants | 6 | 12 | 8 | 2 | 21

3. Primary Outcome: Overall Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) Response Rate Based on Blinded Independent Central Radiology (BICR) Review (Cohorts A, B, C, and D)
Description: Overall Response Rate (ORR) was defined as the percentage of participants who experienced a Complete Response (CR; disappearance of all target lesions) or a Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 based on BICR evaluation. The percentage of participants who experienced a CR or PR for Cohorts A, B, C and D participants was presented for the first course of pembrolizumab treatment per protocol. Cohorts A, B, C and D enrolled participants with programmed cell death-ligand 1 (PD-L1) positive tumors.
Time Frame: Every 8 weeks until disease progression (Cohorts A, B, D: Up to ~ 35 months; Cohort C: Up to ~ 28 months) - through FA cutoff date 26 Apr 2016 (Cohorts: A, B, D) & 01 Sep 2015 (Cohort C)
Population: The population consisted of Cohorts A, B, C and D participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer | Cohort B: Head & Neck Cancer | Cohort C: Urothelial Cancer | Cohort D: Gastric Cancer
Number analyzed (Participants) | 32 | 60 | 33 | 39
Percentage of Participants | 15.6 [5.3 to 32.8] | 16.7 [8.3 to 28.5] | 21.2 [9.0 to 38.9] | 20.5 [9.3 to 36.5]

4. Primary Outcome: Overall RECIST 1.1 Response Rate Based on BICR Review for Participants in Cohort B2
Description: ORR was defined as the percentage of participants in the analysis population who experienced a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 based on BICR evaluation. The percentage of participants who experienced a CR or PR in Cohort B2 was presented for the first course of pembrolizumab treatment per protocol.
Time Frame: Every 8 weeks until disease progression (Up to ~ 35 months) - through FA cutoff date 26 Apr 2016
Population: The population consisted of all Cohort B2 participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort B2: Head & Neck Cancer Expansion
Number analyzed (Participants) | 132
Percentage of Participants | 18.2 [12.0 to 25.8]

5. Secondary Outcome: Overall RECIST 1.1 Response Rate Based on BICR Review, Cohorts B and B2 Human Papilloma Virus (HPV)-Positive Participants
Description: ORR was defined as the percentage of participants in the analysis population who experienced a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 based on BICR evaluation. The percentage of participants who had tumors which were HPV positive and who experienced a CR or PR in the combined Cohorts B2 and B2 was presented for the first course of pembrolizumab treatment per protocol.
Time Frame: Every 8 weeks until disease progression (Up to ~ 35 months) - through FA cutoff date 26 Apr 2016
Population: The population consisted of all Cohort B and Cohort B2 HPV-positive participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohorts B & B2: Head & Neck Cancer HPV-Positive Participants: Participants received pembrolizumab, 10 mg/kg, IV once every 2 weeks or pembrolizumab, 200 mg, IV once every 3 weeks, and continued to receive study drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years). Participants who stopped study treatment without progression (e.g. completed 2 years) may have been eligible for up to 1 year of retreatment upon subsequently experiencing disease progression.
Arm/Group | Cohorts B & B2: Head & Neck Cancer HPV-Positive Participants
Number analyzed (Participants) | 64
Percentage of Participants | 21.9 [12.5 to 34.0]

6. Secondary Outcome: Overall RECIST 1.1 Response Rate Based on BICR Review, Cohort D Asia-Pacific (AP) Participants
Description: ORR was defined as the percentage of participants in the analysis population who experienced a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 based on BICR evaluation. The percentage of participants who were from the Asia Pacific region and experienced a CR or PR in Cohort D was presented for the first course of pembrolizumab treatment per protocol.
Time Frame: Every 8 weeks until disease progression (Up to ~ 35 months) - through FA cutoff date 26 Apr 2016
Population: The population consisted of all Cohort D participants from AP region who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohort D: Gastric Cancer AP Participants: Participants who were from the Asia Pacific region received pembrolizumab, 10 mg/kg, IV once every 2 weeks, and continued to receive study drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years). Participants who stopped study treatment without progression (e.g. completed 2 years) may have been eligible for up to 1 year of retreatment upon subsequently experiencing disease progression.
Arm/Group | Cohort D: Gastric Cancer AP Participants
Number analyzed (Participants) | 19
Percentage of Participants | 21.1 [6.1 to 45.6]

7. Secondary Outcome: Overall RECIST 1.1 Response Rate Based on BICR Review, for Participants Previously Treated With Cetuximab and Platinum in Cohorts B and B2
Description: ORR was defined as the percentage of participants in the analysis population who experienced a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) and was assessed using RECIST 1.1 based on BICR evaluation. The percentage of participants who were previously treated with cetuximab and platinum and experienced a CR or PR in the Cohorts B and B2 was presented for the first course of pembrolizumab treatment per protocol.
Time Frame: Every 8 weeks until disease progression (Up to ~ 35 months) - through FA cutoff date 26 Apr 2016
Population: The population consisted of all Cohort B or B2 participants who progressed following cetuximab and platinum therapy and received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Cohorts B & B2: Head & Neck Cancer: Participants received pembrolizumab, 10 mg/kg, IV once every 2 weeks (Cohort B) or pembrolizumab, 200 mg, IV once every 3 weeks (Cohort B2), and continued to receive study drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years). Participants who stopped study treatment without progression (e.g. completed 2 years) may have been eligible for up to 1 year of retreatment upon subsequently experiencing disease progression.
Arm/Group | Cohorts B & B2: Head & Neck Cancer
Number analyzed (Participants) | 110
Percentage of Participants | 14.5 [8.5 to 22.5]

8. Secondary Outcome: Overall RECIST 1.1 Response Rate Based on Investigator Assessment for Cohorts A, B, C and D
Description: ORR was defined as the percentage of participants in the analysis population who experienced a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) and was assessed by Investigator evaluation. The percentage of participants who experienced a CR or PR in Cohorts A, B, C and D based on investigator assessment was presented for the first course of pembrolizumab treatment per protocol. ORR per RECIST 1.1 based on investigator assessment was presented for Cohort B2 in a separate outcome measure.
Time Frame: as for outcome 3
Population: The population consisted of all Cohort A, B, C and D participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort A: Triple Negative Breast Cancer | Cohort B: Head & Neck Cancer | Cohort C: Urothelial Cancer | Cohort D: Gastric Cancer
Number analyzed (Participants) | 32 | 60 | 33 | 39
Percentage of Participants | 15.6 [5.3 to 32.8] | 16.7 [8.3 to 28.5] | 21.2 [9.0 to 38.9] | 33.3 [19.1 to 50.2]

9. Secondary Outcome: Overall RECIST 1.1 Response Rate Based on Investigator Assessment for Cohort B2
Description: ORR was defined as the percentage of participants in the analysis population who experienced a CR (disappearance of all target lesions) or a PR (at least a 30% decrease in the sum of diameters of target lesions) and was assessed by Investigator evaluation. The percentage of participants who experienced a CR or PR in Cohort B2 based on investigator assessment was presented for the first course of pembrolizumab treatment per protocol. ORR per RECIST 1.1 based on investigator assessment was presented for the other cohorts in a separate outcome measure.
Time Frame: Every 8 weeks until disease progression (Up to ~ 35 months) - through FA cutoff date 26 Apr 2016
Population: The population consisted of all Cohort B2 participants who received ≥1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Cohort B2: Head & Neck Cancer Expansion
Number analyzed (Participants) | 132
Percentage of Participants | 20.5 [13.9 to 28.3]

10. Other Pre Specified Outcome: Number of Participants With Log Fold Change From Baseline in Cytokines (Interleukin 10 [IL-10]) >1
Description: IL-10 is an anti-inflammatory cytokine. The number of participants with a log fold change from Baseline in IL-10 >1 was to be presented. Protocol Amendment 03 (26 May 2015) removed the secondary objective of investigating the relationship between programmed cell death 1 (PD-1) inhibition and up-regulation of cytokines biomarkers predicting response (e.g. IL-10) from the protocol. No data were collected for this outcome measure.
Time Frame: Baseline and Week 8
Population: The population was to consist of all allocated participants who: 1) received ≥1 dose of study treatment and 2) had a baseline IL-10 assessment, and 3) had a post baseline IL-10 assessment. No data were collected for this outcome measure.
Arm/Group | Cohort A: Triple Negative Breast Cancer | Cohort B: Head & Neck Cancer | Cohort C: Urothelial Cancer | Cohort D: Gastric Cancer | Cohort B2: Head & Neck Cancer Expansion
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious and non-serious AEs were collected up to ~ 71 months and all-cause mortality up to ~ 85 months for pembrolizumab first and second course treatment (through end of trial (EOT) cutoff date 30 June 2020).
Description: All-cause mortality was reported on all allocated participants (first and second course). Serious and non-serious AEs were reported among participants who received at least one dose of study treatment. MedDRA preferred terms 'Progressive Disease' and 'Malignant Neoplasm Progression' not related to the drug were excluded.
Groups:
- Cohort A: Triple Negative Breast Cancer; Cohort B: Head & Neck Cancer; Cohort C: Urothelial Cancer; Cohort D: Gastric Cancer: Participants received pembrolizumab, 10 mg/kg, IV once every 2 weeks, and continued to receive study drug until disease progression, death, withdrawal of consent, Investigator decision, or end of study (up to 2 years). Participants who stopped study treatment without progression (e.g. completed 2 years) may have been eligible for up to 1 year of retreatment upon subsequently experiencing disease progression.
Arm/Group | Cohort A: Triple Negative Breast Cancer | Cohort B: Head & Neck Cancer | Cohort C: Urothelial Cancer | Cohort D: Gastric Cancer | Cohort B2: Head & Neck Cancer Expansion
All-Cause Mortality (participants affected / at risk) | 25/32 | 54/61 | 29/33 | 34/39 | 110/132
Serious Adverse Events (participants affected / at risk) | 13/32 | 27/60 | 21/33 | 17/39 | 60/132
Other Adverse Events (participants affected / at risk) | 31/32 | 58/60 | 32/33 | 37/39 | 124/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Triple Negative Breast Cancer (N=32) | Cohort B: Head & Neck Cancer (N=60) | Cohort C: Urothelial Cancer (N=33) | Cohort D: Gastric Cancer (N=39) | Cohort B2: Head & Neck Cancer Expansion (N=132)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Autoimmune colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mouth haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue oedema (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Death (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4)
Face oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fascial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningitis aseptic (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 5 (8) | 1 (1) | 1 (1) | 3 (4)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Streptococcal bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoradionecrosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post lumbar puncture syndrome (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood fibrinogen decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fistula discharge (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to peripheral vascular system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug withdrawal convulsions (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuromyopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pemphigoid (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: Triple Negative Breast Cancer (N=32) | Cohort B: Head & Neck Cancer (N=60) | Cohort C: Urothelial Cancer (N=33) | Cohort D: Gastric Cancer (N=39) | Cohort B2: Head & Neck Cancer Expansion (N=132)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 19 (22) | 7 (7) | 4 (5) | 27 (32)
Lymphopenia (Blood and lymphatic system disorders) | 1 (5) | 5 (6) | 1 (1) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 0 (0) | 2 (10) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 9 (10) | 0 (0) | 5 (5) | 19 (20)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 2 (3)
Abdominal distension (Gastrointestinal disorders) | 3 (3) | 4 (4) | 1 (2) | 3 (3) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 3 (3) | 6 (7) | 13 (16) | 8 (8)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Constipation (Gastrointestinal disorders) | 6 (6) | 15 (17) | 10 (11) | 7 (10) | 21 (22)
Diarrhoea (Gastrointestinal disorders) | 9 (14) | 13 (20) | 3 (3) | 5 (5) | 14 (16)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 6 (7) | 0 (0) | 1 (1) | 16 (16)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 9 (13) | 15 (21) | 9 (12) | 11 (11) | 20 (21)
Oral pain (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 7 (7)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 6 (11)
Vomiting (Gastrointestinal disorders) | 6 (9) | 12 (13) | 6 (8) | 9 (10) | 13 (14)
Asthenia (General disorders) | 1 (1) | 4 (4) | 2 (2) | 3 (3) | 5 (5)
Chest pain (General disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 9 (9)
Chills (General disorders) | 1 (1) | 5 (6) | 3 (4) | 2 (2) | 10 (11)
Face oedema (General disorders) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 1 (1)
Fatigue (General disorders) | 17 (21) | 32 (35) | 17 (19) | 12 (15) | 59 (64)
Malaise (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 7 (7) | 11 (14) | 4 (4) | 7 (8)
Pain (General disorders) | 2 (2) | 4 (4) | 3 (3) | 0 (0) | 5 (5)
Pyrexia (General disorders) | 3 (5) | 12 (15) | 9 (11) | 4 (6) | 22 (25)
Swelling face (General disorders) | 0 (0) | 4 (5) | 0 (0) | 0 (0) | 8 (8)
Temperature intolerance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Candida infection (Infections and infestations) | 1 (1) | 2 (6) | 2 (2) | 0 (0) | 4 (6)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 7 (9)
Pneumonia (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 8 (8)
Sinusitis (Infections and infestations) | 0 (0) | 4 (6) | 3 (3) | 0 (0) | 3 (5)
Skin infection (Infections and infestations) | 0 (0) | 4 (4) | 2 (2) | 0 (0) | 5 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 3 (4) | 2 (3) | 2 (2) | 7 (10)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 6 (8) | 2 (3) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (4) | 2 (3) | 0 (0) | 2 (2) | 3 (3)
Alanine aminotransferase increased (Investigations) | 4 (4) | 2 (3) | 3 (3) | 4 (4) | 6 (7)
Amylase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 2 (3) | 4 (4) | 5 (5) | 8 (10)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 5 (6)
Blood bilirubin increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 4 (4) | 9 (10) | 2 (3) | 4 (4)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (9)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 1 (1) | 10 (10) | 3 (3) | 6 (7) | 25 (32)
Weight increased (Investigations) | 0 (0) | 2 (3) | 3 (4) | 0 (0) | 5 (5)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 14 (14) | 13 (13) | 12 (13) | 30 (31)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 6 (8) | 3 (3) | 0 (0) | 9 (10)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 8 (9)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (11) | 0 (0) | 2 (2) | 6 (6)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 5 (8) | 2 (2) | 1 (1) | 3 (5)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 8 (8)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 11 (25) | 3 (3) | 2 (2) | 10 (11)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 2 (3) | 3 (3) | 8 (9)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 10 (18) | 5 (12) | 2 (2) | 12 (13)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2) | 6 (8) | 2 (4) | 0 (0) | 7 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (12) | 11 (13) | 3 (3) | 6 (6) | 16 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (10) | 6 (7) | 4 (4) | 13 (13)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 3 (3) | 2 (2) | 3 (4)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 1 (2)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (8) | 0 (0) | 0 (0) | 3 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (6) | 2 (2) | 3 (3) | 7 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (12) | 8 (8) | 3 (4) | 3 (3) | 7 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 13 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 3 (3) | 1 (1) | 6 (8)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4) | 2 (2) | 1 (1) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Balance disorder (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 3 (4) | 10 (11) | 2 (2) | 4 (4) | 7 (7)
Headache (Nervous system disorders) | 3 (5) | 10 (12) | 2 (2) | 3 (3) | 13 (15)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 6 (7) | 1 (1) | 0 (0) | 5 (5)
Confusional state (Psychiatric disorders) | 1 (1) | 3 (3) | 4 (4) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 6 (6)
Insomnia (Psychiatric disorders) | 2 (2) | 5 (6) | 0 (0) | 1 (1) | 9 (9)
Restlessness (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 9 (10) | 3 (4) | 8 (9) | 21 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 13 (15) | 7 (7) | 1 (1) | 21 (21)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (10) | 1 (1) | 3 (3) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 2 (2) | 0 (0) | 3 (3)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (7) | 0 (0) | 1 (1) | 6 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 0 (0) | 2 (2) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 12 (14)
Erythema (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (5) | 8 (13) | 3 (4) | 6 (7) | 14 (15)
Rash (Skin and subcutaneous tissue disorders) | 4 (6) | 11 (13) | 2 (2) | 2 (3) | 18 (22)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 7 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Hypotension (Vascular disorders) | 1 (1) | 10 (11) | 3 (3) | 1 (1) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT01848834/Prot_SAP_000.pdf